CLINICAL TRIAL: NCT02131051
Title: Non-interventional Study: Application of Ectoin® Rhinitis Nasal Spray and Eye Drops in Patients With Allergic Rhinitis
Brief Title: Application of Ectoine Containing Nasal Spray and Eye Drops in Patients With Allergic Rhinitis
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: REP-85
Record Dates: First submitted 2014-04-25; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: ectoine; allergic rhinitis; bitop
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Azelastine group: Azelastine nasal spray Azelastine eye drops
- Ectoin group: Ectoin Allergy Nasal Spray Ectoin Allergy Eye Drops

SUMMARY:
This is a comparative, open label, parallel group, non interventional study to further demonstrate the effectiveness and tolerability of Ectoin Allergy Nasal Spray and Eye drops. In addition the effectiveness and safety shall be compared to Azelastine containing nasal Sprays and Eye drops. The patient applied Ectoin® Rhinitis Nasal Spray / Eye drops or takes Azelastine nasals spray and eye drops according to the instructions for use. The observation takes place over a period of 7 days. Response to treatment is recorded at day 7 by the physician and in daily by the patient in a dairy.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* aged 18-70 years
* Patients with proven allergy and acute symptoms in nose and eye which are treated with Ectoin Allergy Nasal Spray and Ectoin Allergy Eye Drops or Azelastine Nasal Spray and Azelastine Eye Drops during the observational period

Exclusion Criteria:

* pregnancy and nursing women,
* drug addicts and persons unable to give consent to study participation,
* patients with intolerance against ingredients of any of the study treatments,
* previous eye or nose surgery,
* concomitant treatment with anti-allergic drugs, and
* diseases which might influence the output of the study according to the physicians' judgment.
* contra indications according to the label

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in primary allergic symptoms symptoms | Day1, Day 7
  Change in the primary allergic nasal and ophthalmic symptoms:
  Degree of nasal breathing impairment, Rhinorrhea, Frequency of sneezing, Nasal itching,Eye itching, Watery eyes, Conjunctivitis score (eye redness)

SECONDARY OUTCOMES:
Palatal itching score | day 1 and day 7
Efficacy and tolerability assessment by the patients | day1 and day 7
  Patients assess the efficacy and tolerability separately based on a general an Scale from 0 to 8

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Sonnemann, MD, Principal Investigator — HNO Praxis Elmshorn
Locations (1):
- HNO Praxis Elmshorn, Elmshorn, Germany